CLINICAL TRIAL: NCT05915780
Title: Effects of Aerobic Exercises on Static & Dynamic Balance in Children With Down's Syndrome
Brief Title: Effect of Aerobic Exercises on Static & Dynamic Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0712
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Down Syndrome
Keywords: Down syndrome; aerobic exercises; Static & dynamic balance
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: It is a randomized control trial, used to compare the effect of aerobic exercises on static & dynamic balance in children with down's syndrome. Subjects with down syndrome meeting the predetermined inclusion & exclusion criteria will be divided into two groups using simple random sampling technique
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols & possible efforts will be put to mask the both groups about their treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will be administered with the cycling exercises in addition to the complete plan of care that is being administered to the control group. The cycling intervention will be performed 3 times per week, for 30 minutes, within a 8-week period
  Interventions: Device: Cycling
- Controlled (Other): Control group will be given with the standard physical therapy intervention that includes progressive resistance training that will be performed using weights, two sets of 10 repetitions will be given for each muscle group, resistance will be increased by ½ Kg as children are able to complete without undue stresses); balance exercises (stand on a balance board, one-leg stance, heal-to-toes stance, walking on balance board, walking on a balance beam, walking on a line, and walking on the inclined surface); flexibility exercises (if required);
  Interventions: Device: Balance Board

INTERVENTIONS:
Device: Cycling — The experimental group will be administered with the cycling exercises in addition to the complete plan of care that is being administered to the control group. The cycling intervention will be performed 3 times per week, for 30 minutes, within a 8-week period
  Arms: Experimental
Device: Balance Board — Control group will be given with the standard physical therapy intervention that includes progressive resistance training that will be performed using weights, two sets of 10 repetitions will be given for each muscle group, resistance will be increased by ½ Kg as children are able to complete without undue stresses); balance exercises (stand on a balance board, one-leg stance, heal-to-toes stance, walking on balance board, walking on a balance beam, walking on a line, and walking on the inclined surface); flexibility exercises (if required);
  Arms: Controlled

SUMMARY:
To determine the effect of aerobic exercises on static & dynamic balance of children in Down syndrome. When a person has Down syndrome, they have an extra chromosome. In the body, chromosomes are discrete collections of genes. They control how a baby's body develops and works both throughout pregnancy and after birth. A newborn typically has 46 chromosomes. Down syndrome is a genetic disorder that affects physical and developmental growth and can cause minor to severe issues. Mental impairment, unusual facial features, an increased risk of cardiac defects, and digestive issues that can range in severity from mild to severe are all symptoms associated with the syndrome.

DETAILED DESCRIPTION:
This will be a randomized controlled trial. Total sample size of 20 will be divided into control and experimental groups. Control group will be given with the standard physical therapy intervention as a baseline treatment while experimental group will be given with the aerobic exercise along with baseline treatment. Pediatric balance test and the six-minute walk test will be used before and after the intervention. Data will be analyzed on SPSS 26.0 and necessary analysis will be done after checking the normality of data.

ELIGIBILITY:
Inclusion Criteria:

* Children with medical diagnosis of DS
* Children with mild (IQ 50-70) to moderate (IQ 35-40) mental retardation
* Age 5-12 Years
* Children who were able to stand and walk

Exclusion Criteria:

* Recent injury to lower extremities
* History of or ongoing vestibular neuritis
* Use of Walking Aids

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg Balance Scale | 8 weeks
  The scale quantifies balance impairments in daily life activities by scoring 0-4 points for the ability to maintain balance while sitting and standing, during 360 degree turns and transfers between juxtaposed chairs, when picking objects from the floor, placing an alternate feet on a stool and leaning forward in a standing position.
Time Up & Go | 8 Weeks
  Time up & go test is a simple test used to assess a person's mobility & requires both static & dynamic balance.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair and sit down while turning 180 degrees Interpretation: ≤ 10 seconds= normal. ≤20 seconds = good mobility, can go out alone, mobile without gait aid. ≤ 30 seconds= problems, cannot go outside alone, requires gait aid. A score of ≥ 14 seconds has been shown to indicate high risk of falls.
6 Minutes Walk Test | 8 weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity Six-Minute Walk Test recommend use of a 30 meter or 100 foot walkway with the length of the corridor marked every 3 meters.

CONTACTS AND LOCATIONS:
Overall Officials: Usman Arif, *MS, Study Chair — Student
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No